CLINICAL TRIAL: NCT05405452
Title: Investigation of the Effectiveness of Vibratory Stimulus in Trigger Finger Injections
Brief Title: Vibratory Anesthesia in Trigger Finger Injections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Tolga Turker, Associate Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001135
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Trigger Finger; Pain; Anesthesia, Local
MeSH Terms: conditions — Trigger Finger Disorder; Pain | interventions — Ethyl Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- No topical anesthesia (No Intervention): No topical anesthesia will be given during the trigger finger injection.
- Topical coolant (Experimental): The subject will have 5 seconds of sterile ethyl chloride sprayed at the site of the trigger finger injections just prior to the administration of the injection.
  Interventions: Drug: Gebauers Ethyl Chloride 100% Topical Spray
- Vibration (Experimental): The subject will have a vibration device placed just proximal to the site of the trigger finger injection concurrent with the administration of the injection.
  Interventions: Device: Vibration Anesthesia Device by Blaine Labs

INTERVENTIONS:
Device: Vibration Anesthesia Device by Blaine Labs — Device which vibrates on top of skin
  Arms: Vibration
Drug: Gebauers Ethyl Chloride 100% Topical Spray — Sterile ethyl chloride spray
  Other Names: P/N 0386-0001-03
  Arms: Topical coolant

SUMMARY:
This study aims to compare the effectiveness of the use of no topical anesthesia, topical coolant, and the use of vibration in the reduction of pain during trigger finger injections. This will be done by randomizing patients who are diagnosed with trigger finger, warrant and choose to continue with a steroid injection into each of the respective anesthetic (or lack thereof) methods described. After conducting this and gathering data on the subjects pain felt, we will compare the analgesia from each of the anesthetic methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult
* Diagnosed with trigger finger
* Warrants a trigger finger injection

Exclusion Criteria:

* Subjects with known decreased light touch sensation in the territory of the trigger finger injection.
* Not diagnosed with trigger finger or does not warrant a trigger finger injection per the typical treatment algorithm adopted by the attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain Felt | Immediately after the trigger finger injection is completed
  Visual Analog Pain Scale Rating (Hayes and Patterson 1921)
  Scale Title: Pain scale Maximum Value: 10 - The worst pain Minimum value: 0 - No pain
  *A lower number indicates a better outcome (less pain felt).

CONTACTS AND LOCATIONS:
Overall Officials: Tolga Turker, MD, Principal Investigator — Associate Professor
Locations (2):
- United States (2):
  - Banner UMC North Hills Clinic, Tucson, Arizona
  - Banner University Alvernon Clinic, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blazar, P. and R. Aggarwal, Trigger finger (stenosing flexor tenosynovitis). 2018.
- [Background] Sampson SP, Badalamente MA, Hurst LC, Seidman J. Pathobiology of the human A1 pulley in trigger finger. J Hand Surg Am. 1991 Jul;16(4):714-21. doi: 10.1016/0363-5023(91)90200-u. PMID 1880372
- [Background] Sbernardori MC, Bandiera P. Histopathology of the A1 pulley in adult trigger fingers. J Hand Surg Eur Vol. 2007 Oct;32(5):556-9. doi: 10.1016/J.JHSE.2007.06.002. Epub 2007 Aug 7. PMID 17950222
- [Background] Makkouk AH, Oetgen ME, Swigart CR, Dodds SD. Trigger finger: etiology, evaluation, and treatment. Curr Rev Musculoskelet Med. 2008 Jun;1(2):92-6. doi: 10.1007/s12178-007-9012-1. PMID 19468879
- [Background] Petchprapa CN, Vaswani D. MRI of the Fingers: An Update. AJR Am J Roentgenol. 2019 Sep;213(3):534-548. doi: 10.2214/AJR.19.21217. Epub 2019 Jul 3. PMID 31268729
- [Background] Lunsford D, Valdes K, Hengy S. Conservative management of trigger finger: A systematic review. J Hand Ther. 2019 Apr-Jun;32(2):212-221. doi: 10.1016/j.jht.2017.10.016. Epub 2017 Dec 28. PMID 29290504
- [Background] Dala-Ali BM, Nakhdjevani A, Lloyd MA, Schreuder FB. The efficacy of steroid injection in the treatment of trigger finger. Clin Orthop Surg. 2012 Dec;4(4):263-8. doi: 10.4055/cios.2012.4.4.263. Epub 2012 Nov 16. PMID 23205235
- [Background] Wojahn RD, Foeger NC, Gelberman RH, Calfee RP. Long-term outcomes following a single corticosteroid injection for trigger finger. J Bone Joint Surg Am. 2014 Nov 19;96(22):1849-54. doi: 10.2106/JBJS.N.00004. PMID 25410501
- [Background] Franko OI, Stern PJ. Use and Effectiveness of Ethyl Chloride for Hand Injections. J Hand Surg Am. 2017 Mar;42(3):175-181.e1. doi: 10.1016/j.jhsa.2016.12.013. PMID 28259274
- [Background] Moayedi M, Davis KD. Theories of pain: from specificity to gate control. J Neurophysiol. 2013 Jan;109(1):5-12. doi: 10.1152/jn.00457.2012. Epub 2012 Oct 3. PMID 23034364
- [Background] Sharma P, Czyz CN, Wulc AE. Investigating the efficacy of vibration anesthesia to reduce pain from cosmetic botulinum toxin injections. Aesthet Surg J. 2011 Nov;31(8):966-71. doi: 10.1177/1090820X11422809. Epub 2011 Oct 14. PMID 22001341
- [Background] Nanitsos E, Vartuli R, Forte A, Dennison PJ, Peck CC. The effect of vibration on pain during local anaesthesia injections. Aust Dent J. 2009 Jun;54(2):94-100. doi: 10.1111/j.1834-7819.2009.01100.x. PMID 19473149
- [Background] Nasehi A, Bhardwaj S, Kamath AT, Gadicherla S, Pentapati KC. Clinical pain evaluation with intraoral vibration device during local anesthetic injections. J Clin Exp Dent. 2015 Feb 1;7(1):e23-7. doi: 10.4317/jced.51643. eCollection 2015 Feb. PMID 25810837
- [Background] Park KY, Lee Y, Hong JY, Chung WS, Kim MN, Kim BJ. Vibration Anesthesia for Pain Reduction During Intralesional Steroid Injection for Keloid Treatment. Dermatol Surg. 2017 May;43(5):724-727. doi: 10.1097/DSS.0000000000001040. PMID 28244902
- [Background] Smith KC, Comite SL, Balasubramanian S, Carver A, Liu JF. Vibration anesthesia: a noninvasive method of reducing discomfort prior to dermatologic procedures. Dermatol Online J. 2004 Oct 15;10(2):1. PMID 15530291